CLINICAL TRIAL: NCT02656849
Title: A Phase II Study of BAY 1000394 in MCL1-Amplified, MYC-Amplified, CCNE1-Amplified Tumors
Brief Title: BAY 1000394 for MCL-1-, MYC-, and CCNE1-Amplified Tumors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Development of BAY1000394 has been terminated by Bayer.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Geoffrey Shapiro, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-380
Record Dates: First submitted 2016-01-11; First posted 2016-01-15 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Solid Tumor
Keywords: Solid Tumor
MeSH Terms: interventions — roniciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BAY 1000394 (Experimental): After the screening procedures confirm eligibility to participate in the research study:
  * Each treatment cycle lasts 4 weeks.
  * Participants will take the study drug orally at predetermined times and dosage per cycle.
  Interventions: Drug: BAY 1000394

INTERVENTIONS:
Drug: BAY 1000394
  Other Names: Roniciclib

SUMMARY:
This research study is studying whether a new experimental cancer study drug BAY 1000394 will be helpful in treating solid tumor cancer with an abnormality in one of the following genes: Mcl-1, Myc or CCNE.

DETAILED DESCRIPTION:
* This research study is a Phase II clinical trial. Phase II clinical trials test the effectiveness of an investigational drug to learn whether the drug works in treating a specific cancer.
* "Investigational" means that the drug is still being studied and that research doctors are trying to find out more about it-such as the safest dose to use, the side effects it may cause, and if the drug is effective for treating different types of cancer.
* It also means that the FDA (the U.S. Food and Drug Administration) has not approved BAY 1000394 for use in participants with your type of cancer.
* The study drug is a pan-CDK inhibitor targeting the genetic defect in several tumors, MCL1, Myc, or CCNE.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have advanced cancer for which no curative therapy exists and have a malignancy which matches one of the following cohorts:

  * MCL1 amplification (≥ 3 fold);
  * MYC amplification (≥ 6 fold);
  * CCNE1 amplification (≥ 6 fold).
  * Molecular abnormalities may be detected by any CLIA-certified test, including Massive Parallel (Next-Generation) sequencing platforms.
* Patients must have measurable disease as defined by RECIST 1.1 criteria. In selected cases patients with evaluable disease may be eligible after discussion between the PI and Bayer.
* Participants must have completed at least one line of therapy in the advanced/metastatic setting prior to enrollment
* Participants with advanced disease for which approved second-line options exist will be eligible when they have progressed beyond such approved second-line therapy
* Age ≥ 18 years. Because there is no data for evaluating these compounds in pediatric populations, the appropriate clinical trial can be conducted in the future in this specific population.
* ECOG performance status of 0-1 (Karnofsky ≥70%, see Appendix A)
* Life expectancy of greater than 12 weeks
* Adequate bone marrow, liver, and renal functions as assessed by the following laboratory requirements:

  * Hemoglobin ≥8.5 g/dL
  * Absolute neutrophil count (ANC) ≥2 x 10/9/L
  * Platelet count ≥100 x 10/9/L
  * Total bilirubin ≤1.5 times the upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤2.5 x ULN (≤5 x ULN for subjects with liver involvement of their cancer)
  * Prothrombin time-international normalized ratio (PT-INR) and partial thromboplastin time (aPTT) ≤1.5 x ULN
  * Estimated glomerular filtration rate (eGFR) ≥60 mL/min per 1.73 m/2 according to the Cockcroft-Gault formula
* Negative serum pregnancy test in women of childbearing potential (WOCBP)(performed within 7 days of randomization). Negative results must be available prior to study treatment administration
* Women of childbearing potential and men must agree to use adequate barrier birth control measures from the time of signing of the informed consent form until at least 3 months after the last study drug administration. The investigator or a designated associate is requested to advise the subject on how to achieve adequate birth control. Adequate contraception is defined in the study as any medically recommended method (or combination of methods) as per standard of care. These procedures should be documented in source documents. Postmenopausal women are defined as:

  * Age >50 years with amenorrhea for at least 12 months or
  * Age ≤50 years with 6 months of spontaneous amenorrhea and follicle stimulating hormone level within postmenopausal range (>40 mIU/mL) or
  * Bilateral oophorectomy
  * Additional adequate contraception which includes hormonal contraception with implants or combined oral contraceptives, certain intrauterine devices, bilateral tubal ligation, hysterectomy, or vasectomy of the partner is allowed as long as a barrier method is also being used
  * Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior radiotherapy is permitted but must have occurred ≥2 weeks (palliative radiotherapy) or ≥ 4 weeks (curative radiotherapy) and subject must have no Grade 3 or 4 toxicities prior to first dose of study treatment
* Prior chemotherapy is allowed. Patients must not have received chemotherapy for 3 weeks prior to the initiation of study treatment and must have full recovery from any acute effects of any prior chemotherapy. Patients must not have had nitrosoureas or mitomycin C for 6 weeks prior to the initiation of study treatment.
* Prior exposure to approved receptor tyrosine kinase inhibitors is permitted. At least 5 half-lives must have elapsed since the completion of the kinase inhibitor and the initiation of study treatment.
* Prior experimental (non-FDA approved) therapies and immunotherapies are allowed. Patients must not have received these therapies for 4 weeks prior to the initiation of study treatment and must have full recovery from any acute effects of these therapies.
* Participants must not have received pan-cyclin-dependent kinase inhibitors as prior therapy.
* Current or ongoing administration of anticoagulation or antiplatelet therapy. However, use of low-dose aspirin (≤100 mg/day) and/or low-dose heparin is permitted unless it is being used for conditions other than cancer
* Known hypersensitivity to any of the study treatments or excipients of the preparations or any agent given in association with this study
* Previous deep vein thrombosis (within the last 6 months), arterial thrombotic events (including strokes), or pulmonary embolism
* History of cardiac disease: Congestive heart failure New York Heart Association (NYHA) Class III or IV angina (within past 6 months prior to study entry), myocardial infarction, or cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* Known human immunodeficiency virus infection, active hepatitis B or C, or chronic hepatitis B or C requiring treatment with antiviral therapy
* Active clinically serious infections of NCI-CTCAE v4.0 >Grade 2
* Seizure disorder requiring therapy (such as steroids or anti-epileptics)
* Concomitant use of other medications that are known to lower the seizure threshold
* Symptomatic metastatic brain or meningeal tumors, including those of the spinal cord, and including cases of neoplastic meningitis (also known as carcinomatous meningitis or leptomeningeal carcinomatosis).
* History of organ allograft
* Evidence or history of bleeding disorder, i.e. any hemorrhage / bleeding event of NCI-CTCAE v4.0 >Grade 2 within 4 weeks prior to the first dose of study treatment
* Uncontrolled hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure >90 mmHg despite optimal medical management)
* Serious, non-healing wound, ulcer, or bone fracture (bone fractures due to bone metastases are acceptable)
* Subjects on dialysis
* Sensory neuropathy with sensory alterations or paresthesia (including tingling), interfering with function (≥NCI-CTCAE v4.0 Grade 2)
* Previous or coexisting cancer that is distinct from the study indication and has not been curatively treated >3 years prior to study entry EXCEPT cervical cancer in-situ, treated basal cell carcinoma, superficial bladder tumors (Ta and Tis)
* Any condition that is unstable or could jeopardize the safety of the subject and his/her compliance in the study
* Subjects unable to swallow oral medications
* Any malabsorption condition
* Major surgery, open biopsy, or significant trauma within 4 weeks prior to the first dose of study treatment is excluded (central line surgery is not considered major surgery)
* Autologous bone marrow transplant or stem cell rescue within 4 months prior to first dose of study treatment is not allowed
* Investigational drug treatment outside of this study during or within 4 weeks prior to study entry. Toxic effects of previous investigational drug treatment have to be normalized
* Potent CYP3A4 inhibitors and CYP3A inducers (see Appendix B)
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2019-10 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Six-month progression-free survival rate | six months
  RECIST 1.1

SECONDARY OUTCOMES:
Response Rate Mcl1-amplified tumors | six months
  RECIST 1.1
Response Rate MYC-amplified tumors | six months
  RECIST 1.1
Response Rate CCNE1-amplified tumors | six months
  RECIST 1.1
Overall Survival | six months
  Kaplan Meier analysis
Time to Progression | six months
  RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Shapiro, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States